CLINICAL TRIAL: NCT03906656
Title: Multinational Randomized Controlled Cross-over Trial Comparing C -Brace to Conventional Knee Ankle Foot Orthoses With Respect to Balance, Fall Risk and Activities of Daily Living
Brief Title: Clinical Trial Comparing C-Brace to Knee Ankle Foot Orthosis (KAFO)/Stance Control Orthosis (SCO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PS00120016A-001
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Pareses, Lower Extremity
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Intervention Model Description: Prospective international multi-center, open-labeled randomized, controlled cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KAFO/SCO (Active Comparator): Home use of 3 months with existing knee ankle foot orthosis (KAFO) or existing stance control orthosis (SCO)
  Interventions: Device: KAFO/SCO
- C-Brace (Experimental): Home use of 3 months with newly fitted C-Brace microprocessor-controlled stance and swing control orthosis.
  Interventions: Device: C-Brace

INTERVENTIONS:
Device: C-Brace — The C-Brace consists of individually fabricated thigh, calf and foot components. An ankle joint, unilateral or bilateral fitting, or an individual spring element connects the foot and calf components. The sensor system continuously measures the flexion of the knee joint and its angular acceleration. This allows the C-Brace to detect the user's current walking phase, so it can regulate the hydraulic resistances as well as control the flexion and extension of the knee joint.
  Other Names: Microprocessor-controlled Stance and Swing Orthosis (MP-SSCO)
  Arms: C-Brace
Device: KAFO/SCO — Current knee ankle foot orthosis that the subject was wearing at baseline
  Other Names: Locked KAFO, Posterior offset KAFO, Stance Control Orthosis
  Arms: KAFO/SCO

SUMMARY:
Prospective, international, multi-center, open-labeled, randomized, controlled cross-over trial to evaluate effectiveness and benefits in patients with lower limb impairment in activities of daily living comparing the C-Brace microprocessor-controlled stance and swing orthosis to standard of care use of knee ankle foot orthosis/stance control orthoses

DETAILED DESCRIPTION:
After obtaining informed consent, patients will be screened. For subjects fulfilling inclusion/exclusion criteria, a first baseline assessment will be conducted. Within one to two days, a second set of baseline data will be collected for performance measures. Subjects will then be randomly assigned to be fitted with C-Brace or to continue wearing the current KAFO/SCO. After fitting, an accommodation period follows that will last up to 14 days prior to the initial home use. The first follow-up data collection will occur after three months of the initial home use period. Afterwards, the patients will cross over to KAFO/SCO or C-Brace, respectively. The participants who were fitted with C-Brace will cross over to KAFO/SCO and vice versa. Another accommodation phase will be offered for both C-Brace and KAFO/SCO wearers to ensure that subjects can properly use both devices before the cross-over home use period. The second follow-up data collection will occur after 3-months of the cross-over home use period. At the end of the study, the patients can choose to keep the C-Brace for up to 24 months until reimbursement or to return to their original KAFO/SCO.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been tested with the Trial Tool (DTO) and demonstrated the potential to utilize the C-Brace successfully
* Patient has a BBS score < 45
* Lower limb functional impairment according to CE label wording
* Prior active and compliant use of unilateral or bilateral KAFO or SCO in the past 3 months prior to enrollment in the study
* Patient meets minimum physical requirements to be fitted with a C-Brace, such as muscle status, joint mobility, leg axis and proper control of the orthosis must be guaranteed.
* The User must fulfill the physical and mental requirements for perceiving optical/acoustic signals and/or mechanical vibrations
* The existing muscle strength of the hip extensors and flexors must permit the controlled swing-through of the limb (compensation using the hip is possible).
* Patient´s commitment to use C-Brace 2 at least 1-2 hours per day 5 days per week-
* Patient is ≥ 18 years old
* Patient is willing and able to independently provide informed consent.
* Person is willing to comply with study procedures

Exclusion Criteria:

* Patient who is not able to follow the entire study visits or is unwilling/unable to follow the instructions
* Patient was not able to use DTO
* Patient who is not using an orthosis at least 1 to 2 hours/ day for 5 days per week
* Patient with body weight > 125 kg (includes body weight and heaviest object (weight) carried)
* Patient with Orthoprosthesis
* Patient with flexion contracture in the knee and/or hip joint in excess of 10°
* Patient with uncontrolled moderate to severe spasticity (relative contraindication moderate spasticity)
* Leg length discrepancy in excess of 15 cm
* Patient with unstable neurological or cardiovascular/pulmonary disease, cancer
* Pregnancy
* Patient using a C-Brace
* Patient with known vertigo or with history of falls unrelated to orthosis use or unrelated to motor disability
* Patient who has never been fitted an orthosis before
* Patient is not able to answer the self-administered questionnaires independently; for patients with upper extremity impairment is it allowed to verbally answer the questions.
* Patient participating already in a study during this study´s duration
* Patient participated in earlier C-Brace studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Braatz, Dr. med., Principal Investigator — Zentrum für Healthcare Technology der Privaten Hochschule Göttingen
Locations (13):
- United States (4):
  - Hanger Clinic, Sarasota, Florida
  - Scheck & Siress, Chicago, Illinois
  - Hanger Clinic, Houston, Texas
  - Hanger Clinic, Seattle, Washington
- Orthopädisches Spital Speising Speisingerstraße 109, Vienna, Austria
- Germany (7):
  - BeMoveD - Berlin Movement Diagnostics, Berlin, Deutschland
  - Katholisches Klinikum Koblenz-Montabaur, Koblenz, Rhineland-Palatinate
  - Johannesbad Raupennest GmbH & Co. KG, Altenberg
  - Zentrum für Healthcare Technology der Privaten Hochschule Göttingen, Göttingen
  - BG Klinikum Hamburg gGmbH Zentrum für Rehabilitationsmedizin, Hamburg
  - Universitätsklinikum Heidelberg, Zentrum für Orthopädie, Unfallchirurgie und Paraplegiologie, Heidelberg
  - Pohlig GmbH, Traunstein
- Adelante Kenniscentrum, Hoensbroek, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were pre-screened based on their medical and/or orthotic records. After signing a written informed consent, participants were screened for inclusion and exclusion criteria. The screening process comprised a thorough patient evaluation and a test with the functional C-Brace trial tool to check whether the potential study participant was able to initiate swing and utilize controlled knee flexion during weight bearing.
Pre-assignment Details: 149 subjects were enrolled, and 41 failed screening (27 due to BBS score above 44, 11 failed the C-Brace trial tool assessment, 1 had a contraindication for the C-Brace, 1 had a history of vertigo, and 1 was geographically inaccessible). In addition, another 6 subjects dropped out after screening, but prior to randomization. Reasons for these early dropouts were lack of time (2) and personal problems (1) resulting in 102 patients randomized.
Groups:
- KAFO/SCO, Then C-Brace: Home use of 3 months with existing knee ankle foot orthosis (KAFO) or existing stance control orthosis (SCO)
  KAFO/SCO: Current knee ankle foot orthosis that the subject was wearing at baseline
  Crossover immediately after first home-use period to being fit with C-Brace, receiving training, and starting 3-month home-use period as soon as the subject demonstrates he/she is able to use it safely.
- C-Brace, Then KAFO/SCO: Home use of 3 months with newly fitted C-Brace microprocessor-controlled stance and swing control orthosis.
  C-Brace: The C-Brace consists of individually fabricated thigh, calf and foot components. An ankle joint, unilateral or bilateral fitting, or an individual spring element connects the foot and calf components. The sensor system continuously measures the flexion of the knee joint and its angular acceleration. This allows the C-Brace to detect the user's current walking phase, so it can regulate the hydraulic resistances as well as control the flexion and extension of the knee joint.
  Crossover to wearing previous KAFO/SCO, receives training if necessary, wears KAFO/SCO for a 1-month washout period then starting 3-month KAFO/SCO home-use period.
Period: Fitting/Assessment Prior to Home Use 1
Arm/Group | KAFO/SCO, Then C-Brace | C-Brace, Then KAFO/SCO
Started | 52 | 50
Completed | 50 | 47
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Lack of access to site during COVID | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Home Use 1 (3 Months)
Arm/Group | KAFO/SCO, Then C-Brace | C-Brace, Then KAFO/SCO
Started | 50 | 47
Completed | 47 | 44
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 0
Period: Fitting/Assessment Prior to Home Use 2
Arm/Group | KAFO/SCO, Then C-Brace | C-Brace, Then KAFO/SCO
Started | 47 | 44
Completed | 41 | 43
Not Completed | 6 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Lack of access to site during COVID | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Personal problems | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Home Use 2 (3 Months)
Arm/Group | KAFO/SCO, Then C-Brace | C-Brace, Then KAFO/SCO
Started | 41 | 43
Completed | 35 | 41
Not Completed | 6 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Could not cope with KAFO after C-Brace | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat Group
Groups:
- Total: Total of all reporting groups
Arm/Group | KAFO/SCO, Then C-Brace | C-Brace, Then KAFO/SCO | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (15.2) | 55.4 (12.4) | 55.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 26 | 31 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 40 | 38 | 78
  Asian | 6 | 6 | 12
  Black or African American | 2 | 2 | 4
  Other | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Netherlands | 4 | 3 | 7
  Austria | 0 | 1 | 1
  United States | 20 | 22 | 42
  Germany | 28 | 24 | 52
Body Weight [Mean (Standard Deviation); unit: kg] | 77.5 (15.8) | 82.8 (16.3) | 80.1 (16.2)
Height [Mean (Standard Deviation); unit: cm] | 170.1 (11.3) | 170.3 (11.3) | 170.2 (11.2)
Work/employment status [Count of Participants; unit: Participants]
  Employed | 17 | 25 | 42
  Retired | 22 | 21 | 43
  Unemployed | 13 | 4 | 17
Side/bilateral orthosis [Count of Participants; unit: Participants]
  Right | 18 | 23 | 41
  Left | 26 | 21 | 47
  Bilateral | 8 | 6 | 14
Type of orthosis used before study and as control [Number; unit: participants] — This includes bilateral patients, so the number of orthoses will exceed the total number of participants
  participants
    Locked KAFO | 22 | 23 | 45
    Posterior-offset KAFO | 15 | 14 | 29
    SCO (electrical) | 9 | 5 | 14
    SCO (mechanical) | 11 | 13 | 24
    Other | 1 | 1 | 2
Use of walking aids inside [Count of Participants; unit: Participants] — Did the participant use walking aids indoors? Population: Missing data for one patient
  Participants
    number analyzed (Participants) | 51 | 50 | 101
    Yes | 31 | 30 | 61
    No | 20 | 20 | 40
Use of walking aids outside [Count of Participants; unit: Participants] — Did the participant use walking aids outdoors? Population: Missing data for one patient
  Participants
    number analyzed (Participants) | 51 | 50 | 101
    Yes | 44 | 42 | 86
    No | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy: Berg Balance Scale (BBS)
Description: The Berg Balance Scale is a 14-item scale designed to measure static and dynamic balance in adults in a clinical setting. The range in score for the BBS is 0 to 56, with higher scores indicating better balance. Points for each item are deducted if the time or distance requirements are not met, the patient's performance requires supervision, or the patient requires assistance from support or examiner.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline measure with currently worn knee ankle foot orthosis (KAFO) or stance control orthosis (SCO)
- KAFO: Measure at end of 3-month home use period with existing knee ankle foot orthosis (KAFO) or existing stance control orthosis (SCO)
- C-Brace: Measure at the end of the 3-month home-use period with newly fitted C-Brace microprocessor-controlled stance and swing control orthosis.
  C-Brace: The C-Brace consists of individually fabricated thigh, calf and foot components. An ankle joint, unilateral or bilateral fitting, or an individual spring element connects the foot and calf components. The sensor system continuously measures the flexion of the knee joint and its angular acceleration. This allows the C-Brace to detect the user's current walking phase, so it can regulate the hydraulic resistances as well as control the flexion and extension of the knee joint.
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 102 | 86 | 77
score on a scale | 33.6 (11.0) | 37.3 (10.5) | 42.0 (9.1)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the mean difference (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.0002, t-test, 2 sided — Adjusted p-values based on Holm-Bonferroni method. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 3.5, Standard Deviation 8.1 — Mean difference is for paired data (n=73). This explains the discrepancy between the mean difference and the difference between the KAFO and C-Brace means (n=86 and n=77, respectively)
Statistical Analysis 2: Comparison: Baseline vs C-Brace; H0: the mean difference (C-Brace - Baseline) <= 0; Test type: Superiority; p < 0.00001, t-test, 2 sided — Adjusted p-values based on Holm-Bonferroni method. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 6.8, Standard Deviation 9.7 — Mean difference is for paired data (n=77). This explains the discrepancy between the mean difference and the difference between the KAFO and C-Brace means (n=86 and n=77, respectively)
Statistical Analysis 3: Comparison: Baseline vs KAFO; KAFO vs. Baseline -- H0: the mean difference (KAFO - Baseline) <= 0; Test type: Superiority; p < 0.00001, t-test, 2 sided; Mean Difference (Final Values) = 3.3, Standard Deviation 6.3 — Mean difference is for paired data (n=86). This explains the discrepancy between the mean difference and the difference between the Baseline and KAFO means (n=102 and n=86, respectively)

2. Secondary Outcome: Activity-specific Balance Confidence (ABC) Scale
Description: Assessment of patient-perceived balance confidence for 16 activities of daily living. For each activity, subjects rate their level of confidence in doing the activity without losing their balance or becoming unsteady on a scale from 0% to 100%, with 100% being the highest level of confidence. The total score for the ABC scale is an average of all activity scores.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 96 | 81 | 77
score on a scale | 53.1 (19.2) | 51.0 (18.3) | 62.3 (19.5)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the mean difference (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.005, t-test, 2 sided — P-value not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; 63.6 degrees of freedom; Mean Difference (Final Values) = 7.05, Standard Deviation 26.3

3. Secondary Outcome: Dynamic Gait Index (DGI)
Description: An 8-item test used to assess balance during walking tasks. It has a maximum score of 24 with each item being scored 0-3. A higher score indicates greater balance, and subjects lose a a point on all items for which an assistive device is needed.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 99 | 84 | 77
score on a scale | 12.3 (3.3) | 13.4 (3.2) | 15.7 (3.3)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the mean difference (C-Brace - KAFO) <= 0; Test type: Superiority — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; p = 0.005, t-test, 2 sided — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; 74.4 degrees of freedom; Mean Difference (Final Values) = 1.0, Standard Deviation 3.7

4. Secondary Outcome: 6-minute Walk Test
Description: Distance walked in 6 minutes over 12-meter back-and-forth pathway as a measure of functional exercise capacity.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 101 | 86 | 77
meters | 204.9 (73.9) | 213.7 (80.9) | 226.0 (84.3)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the median of the population differences (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.583, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 0.185, Standard Deviation 53.6; Wilcoxon Signed Rank Test. V=1207.5, effect size r = 0.026, p=0.583

5. Secondary Outcome: Stair Assessment Index (SAI) - Down
Description: A 14-point ordinal scale (0 - 13) used to assess different gait patterns during descent of stairs. The range of total scores for the SAI is from 0 to 26, with a higher score indicating a more normative gait pattern and needing less assistance.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 99 | 86 | 76
score on a scale | 4 (3.3) | 4.5 (3.5) | 6 (4.2)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the median of the population differences (C-Brace - KAFO) <= 0. (SAI - Down); Test type: Superiority; p = 0.0078, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 1.28, Standard Deviation 4.37; Wilcoxon Signed Rank Test V=438, effect size r = 0.21, p=0.008

6. Secondary Outcome: Frequency of Falling
Description: Frequency of falling by using C-Brace compared to KAFO/SCO as measured by the number of falls in 3-month period by recollection at baseline and recorded in a Falls Diary during home-use periods
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: number of falls in a three month period
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 101 | 87 | 79
number of falls in a three month period | 4.9 (20.1) | 4.0 (16.8) | 1.1 (3.3)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; Test type: Superiority; p = 0.0020, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = -3.41, Standard Deviation 17.0; Wilcoxon Signed Rank Test V=267, effect size r = 0.32, p=0.002

7. Secondary Outcome: Fear of Falling
Description: Two questions on patients' fear of falling indoors and outdoors based on an 11-point scale (0 = no fear, 10 = max. fear). The total score will range from 0 to 20, with 20 being maximum fear of falling.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 100 | 86 | 78
score on a scale
  Fear of falling indoors | 3.3 (2.9) | 3.3 (2.8) | 2.2 (2.6)
  Fear of falling outdoors | 5.5 (3.0) | 5.2 (2.9) | 4.4 (3.0)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the median of the population differences (C-Brace - KAFO) <= 0. (Fear of falling - indoors); Test type: Superiority; p = 0.0023, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = -1.11, Standard Deviation 3.178; Wilcoxon Signed Rank Test V=433, effect size r = 0.33, p=0.002
Statistical Analysis 2: Comparison: KAFO vs C-Brace; Test type: Superiority; p = 0.0066, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = -0.973, Standard Deviation 3.43; Wilcoxon Signed Rank Test V=557.5, effect size r = 0.265, p=0.0066

8. Secondary Outcome: Probability of Falling More Than Once When Using C-Brace Compared to KAFO/SCO
Description: Proportion of subjects having reported falling more than once will be compared between KAFO and C-Brace home-use periods
Time Frame: 3 months after initial home use period, and 3 months after cross-over home use period
Population: Paired data including subjects with fall history after both KAFO and C-Brace home use periods
Measure: Count of Participants; unit: Participants
Arm/Group | KAFO | C-Brace
Number analyzed (Participants) | 75 | 75
Participants | 25 | 12
Statistical Analysis 1: Comparison: KAFO vs C-Brace; Paired dataset. H0: The probability of fallers wearing C-Brace becoming non-fallers wearing KAFO is the same as the probability of non-fallers wearing C-Brace becoming fallers wearing KAFO; Test type: Superiority; p = 0.006, McNemar — P-value not adjusted for multiple comparisons

9. Secondary Outcome: Reintegration to Normal Living (RNL) Index Questionnaire
Description: 11 items measuring satisfaction regarding perceived physical functioning, and social and emotional life. Higher scores represent higher levels of participation. The range of the adjusted total score is 0 to 100.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 100 | 86 | 76
score on a scale | 71.5 (19.8) | 71.7 (17.6) | 74.0 (19.8)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the median of the population differences (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.08, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 2.82, Standard Deviation 16.4; Wilcoxon Signed Rank Test. V=1325.5, effect size r = 0.181, p=0.08

10. Secondary Outcome: EQ-5D-5L
Description: Measure of health status composed of 5 dimensions: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, anxiety and depression. Each dimension is rated on a 5-point scale indicating the level of perceived problems for each dimension (level 1 indicating no problems and level 5 indicating extreme problems). The raw score is then aggregated and normalized based on region to a 0 to 1 scale (where 0 represents maximum issues and 1 represents no problems).
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 99 | 88 | 75
score on a scale | 0.71 (0.19) | 0.72 (0.19) | 0.74 (0.18)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; H0: the median of the population differences (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.151, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 0.009, Standard Deviation 0.184 — Wilcoxon Signed Rank Test V=1124.5, effect size r = 0.125 p=0.151

11. Secondary Outcome: Work Limitations Questionnaires WLQ-25
Description: 25-item questionnaire to evaluate at-work disability and productivity loss under four sub-scales: time demands, physical demands, mental/interpersonal demands, and output demands. Scale scores range from 0 (limited none of the time) to 100 (limited all of the time).
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: Intention to Treat Group. If one or more items in a subscale were not answered, the patient was excluded from the analysis of that particular subscale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 38 | 34 | 30
score on a scale
  Mental/Interpersonal: number analyzed (Participants) | 37 | 34 | 30
  Mental/Interpersonal | 86.1 (13.3) | 88.4 (11.5) | 91.0 (13.7)
  Output: number analyzed (Participants) | 37 | 34 | 30
  Output | 82.0 (17.9) | 81.9 (17.0) | 84.6 (17.3)
  Physical: number analyzed (Participants) | 37 | 34 | 30
  Physical | 37.5 (24.8) | 34.5 (23.3) | 24.3 (18.8)
  Time | 79.2 (20.1) | 78.3 (24.6) | 79.8 (19.8)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; WLQ-25 - Physical; Test type: Superiority — H0: the mean of the population differences (C-Brace - KAFO) >= 0; p = 0.281, t-test, 2 sided — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; 16.7 degrees of freedom; Mean Difference (Final Values) = -2.10, Standard Deviation 21.5

12. Secondary Outcome: Orthotics & Prosthetics User Survey (OPUS)
Description: A self-report questionnaire designed to evaluate the outcome of orthotic and prosthetic services. Three of the five domains will be administered: lower extremity functional status (20 items, score ranges from 0 - 80, with high score being easier), health-related quality of life index (23 items, score ranges from 0 - 92, with higher score being better) and satisfaction with device (11 items, score ranges from 11 - 55, with higher score being more satisfaction) scales. The domains of upper limb functional measure and satisfaction with service are not applicable in this study.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 99 | 86 | 77
score on a scale
  Quality of Life: number analyzed (Participants) | 98 | 84 | 77
  Quality of Life | 56.6 (7.3) | 56.9 (6.9) | 58.0 (8.0)
  Lower Extremity Functional Status: number analyzed (Participants) | 99 | 86 | 76
  Lower Extremity Functional Status | 45.3 (6.2) | 46.6 (6.3) | 48.8 (6.3)
  Satisfaction with Device: number analyzed (Participants) | 99 | 86 | 76
  Satisfaction with Device | 49.8 (10.5) | 50.6 (9.7) | 51.3 (13.7)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; OPUS - Low Extremity Functional Status. H0: the mean difference (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.00019, t-test, 2 sided — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; 48.4 degrees of freedom; Mean Difference (Final Values) = 1.99, Standard Deviation 5.18

13. Secondary Outcome: Medical Outcomes Study Short Form (SF-36)
Description: 36-item scale constructed to survey health status and quality of life. It assesses eight health concept scales: physical functioning, role functioning/physical, role functioning/emotional, energy/fatigue, emotional well-being, social functioning, pain and general health. Each scale score ranges from 0 to 100 with 100 being the highest (better) score.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 99 | 88 | 77
score on a scale
  Emotional Wellbeing | 76.2 (16.4) | 75.5 (16.3) | 79.2 (15.16)
  Energy/Fatigue | 52.2 (21.3) | 52.3 (20.3) | 56.8 (20.1)
  General Health | 54.1 (22.2) | 54.2 (23.8) | 58.2 (23.8)
  Health Change | 47.4 (24.2) | 48.0 (26.0) | 56.5 (26.4)
  Pain | 55.6 (25.3) | 57.4 (24.9) | 59.5 (26.7)
  Physical Functioning: number analyzed (Participants) | 98 | 88 | 76
  Physical Functioning | 29.7 (22.6) | 31.1 (23.8) | 44.3 (23.3)
  Role limitations due to emotional problems | 78.1 (36.9) | 82.2 (34.3) | 86.1 (28.8)
  Role limitations due to physical health: number analyzed (Participants) | 98 | 88 | 77
  Role limitations due to physical health | 36.5 (39.7) | 44.9 (43.2) | 51.0 (41.2)
  Social Functioning: number analyzed (Participants) | 98 | 85 | 77
  Social Functioning | 74.2 (23.0) | 75.1 (25.0) | 77.3 (24.4)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; Emotional well-being. H0: the mean difference (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.0226, t-test, 2 sided — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; 22.1 degrees of freedom; Mean Difference (Final Values) = 3.19, Standard Deviation 15.0
Statistical Analysis 2: Comparison: KAFO vs C-Brace; Energy/Fatigue. H0: the mean difference (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.0020, t-test, 2 sided — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 6.79, Standard Deviation 21.1
Statistical Analysis 3: Comparison: KAFO vs C-Brace; Health change. H0: the median of the population differences (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.0049, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 10.1, Standard Deviation 29.528; Wilcoxon Signed Rank Test. V=649, effect size r = 0.285, p=0.00493
Statistical Analysis 4: Comparison: KAFO vs C-Brace; Physical Functioning Score. H0: the mean difference (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.0000647, t-test, 2 sided — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; 37.35 degrees of freedom; Mean Difference (Final Values) = 12.6, Standard Deviation 29.2

14. Secondary Outcome: Quebec User Evaluation on Satisfaction With Assistive Technology (QUEST)
Description: 12-item instrument used to assess satisfaction with a specific assistive device. Each questions is rated on a 5-point scale, with 1=not satisfied at all and 5=very satisfied. The first 8 questions comprise the Device subscale and the last 4, the Services subscale. Each subscale and the total score are presented as averages ranging from 1 to 5, with higher scores representing greater satisfaction.
Time Frame: Baseline, 3 months after initial home use period, and 3 months after cross-over home use period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | KAFO | C-Brace
Number analyzed (Participants) | 98 | 87 | 76
score on a scale
  Device | 4.05 (0.67) | 4.05 (0.72) | 4.00 (0.63)
  Service: number analyzed (Participants) | 98 | 87 | 75
  Service | 4.60 (0.64) | 4.66 (0.70) | 4.79 (0.42)
  Total: number analyzed (Participants) | 98 | 87 | 75
  Total | 4.23 (0.59) | 4.27 (0.64) | 4.27 (0.49)
Statistical Analysis 1: Comparison: KAFO vs C-Brace; Device. H0: the median of the population differences (C-Brace - KAFO) <= 0; Test type: Superiority; p = 0.301, Wilcoxon Signed Rank Test — P-values not adjusted for multiple comparisons. P-values < 0.05 used as threshold for statistical significance; Mean Difference (Final Values) = 0.28, Standard Deviation 0.843; Wilcoxon Signed Rank Test V=1018.5, effect size r = 0.056, p=0.301

15. Secondary Outcome: Patient-Related Outcome Questions
Description: Two questions asking how the specific orthoses affected activities they enjoy and their quality of life. Each question is on a 5-point scale, with 1=much worse and 5=much better.
Time Frame: 3 months after cross-over home use period
Population: Subjects that answered the patient-reported outcome questions after having completed home-use periods with both KAFO/SCO and C-Brace (at Visit 2). 75 subjects provided answers to these questions.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | KAFO/SCO, Then C-Brace | C-Brace, Then KAFO/SCO
Number analyzed (Participants) | 35 | 40
units on a scale
  To what extent has the C-Brace enabled you to engage in the activities that you enjoy? | 4 [3 to 4] | 4 [3.75 to 5]
  To what extent has the C-Brace impacted your quality of life? | 4 [3 to 4.5] | 4 [4 to 5]

ADVERSE EVENTS:
Time Frame: For C-Brace, the period of time for adverse events was the 3-month window after the device had been fitted. In addition to the 3-month home use period, for KAFO/SCO there was often an extra month or two, especially for patients randomized to start with C-Brace since it takes time to fabricate the device and adverse events can occur during that waiting period.
Description: For patients with frequent falls or stumbles, an increase in frequency was considered an adverse event and any falls that resulted in an injury were noted individually as adverse events. Seriousness was determined by the consequences of the event as defined in ISO 14155.
Groups:
- KAFO/SCO: Home use of 3 months with existing knee ankle foot orthosis (KAFO) or existing stance control orthosis (SCO). May also include a period of time when the C-Brace was being fabricated prior to the C-Brace home use of 3 months.
  KAFO/SCO: Current knee ankle foot orthosis that the subject was wearing at baseline
Arm/Group | KAFO/SCO | C-Brace
All-Cause Mortality (participants affected / at risk) | 0/102 | 2/88
Serious Adverse Events (participants affected / at risk) | 10/102 | 6/88
Other Adverse Events (participants affected / at risk) | 66/102 | 57/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | KAFO/SCO (N=102) | C-Brace (N=88)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Cholecystolithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Prostate cancer (Reproductive system and breast disorders) | 0/57 (0) | 1/46 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Systemic scleroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | KAFO/SCO (N=102) | C-Brace (N=88)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased fall frequency (General disorders) | 6 (7) | 1 (1) — A significant increase in falls when comparing one home use period to another
Swelling of legs (General disorders) | 1 (1) | 0 (0)
Cystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Immunodeficiency syndromes (Immune system disorders) | 1 (1) | 0 (0)
Multiple sclerosis aggravated (Immune system disorders) | 2 (2) | 1 (1)
Psoriasis (Immune system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 4 (5)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cold symptoms (Infections and infestations) | 5 (5) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella Infection (Infections and infestations) | 0 (0) | 1 (1)
Stomach Virus (Infections and infestations) | 3 (3) | 1 (1)
Injurious Fall (Injury, poisoning and procedural complications) | 21 (37) | 10 (15) — A complete fall, all the way to the ground, that resulted in an injury
Open Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (7)
Fibula Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in foot (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (7)
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in leg (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (9)
Pain in toe (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Patella Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post polio syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Nervous system disorders) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Additional strap necessary (Product Issues) | 0 (0) | 1 (1)
Alignment Issue (Product Issues) | 0 (0) | 2 (2) — A mismatch between the alignment of the orthosis and the subject's physiologic limb
Battery holder defect (Product Issues) | 1/2 (1) | 0/0 (0)
Beeping (Product Issues) | 1/2 (1) | 3 (3)
Bluetooth Malfunction (Product Issues) | 0/2 (0) | 3 (3) — Connectivity issues to the orthosis via the phone app
Broken Spring (Product Issues) | 4 (4) | 0 (0)
Broken Strap (Product Issues) | 3 (3) | 3 (4)
Broken foot stirrup (Product Issues) | 1 (1) | 0 (0)
Charging Malfunction (Product Issues) | 0/2 (0) | 4 (4)
Clicking/cracking noises (Product Issues) | 0 (0) | 2 (2)
Delamination (Product Issues) | 0 (0) | 1 (1)
Foot plate fracture (Product Issues) | 1 (1) | 2 (2)
Insufficient Padding (Product Issues) | 0 (0) | 1 (1)
Joint Malfunction (Product Issues) | 7 (7) | 2 (3)
Loose Screw (Product Issues) | 4 (5) | 1 (1)
Loss of oil (Product Issues) | 0/2 (0) | 1 (1)
Modified foot plate (Product Issues) | 1 (1) | 0 (0)
Poor Fit (Product Issues) | 1 (1) | 0 (0)
Service Light (Product Issues) | 0/2 (0) | 3 (3)
Unexpected mode switch (Product Issues) | 1/7 (1) | 4 (4) — Either switching to a freeze/safety mode, or free swing unexpectedly
Vaginal bleeding (Reproductive system and breast disorders) | 1/45 (1) | 0/42 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (9)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Epistaxis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was affected by the COVID pandemic. Home-use periods interrupted by the pandemic were restarted, and the study was re-opened for enrollment of another 59 subjects. Neither the subjects nor investigators were blinded for interventions. Only subjects with impaired balance (BBS<45) were included. It is unclear whether the amount of device training was sufficient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03906656/Prot_SAP_000.pdf